CLINICAL TRIAL: NCT00803114
Title: Epidural Morphine Following Vaginal Delivery: A Randomised, Double-Blind, Placebo-Controlled Trial
Brief Title: Epidural Morphine Following Vaginal Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Alison Macarthur, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSHREB 01-0227-A
Record Dates: First submitted 2008-11-07; First posted 2008-12-05 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2008-12

CONDITIONS: Pain
Keywords: Postpartum perineal pain; Epidural morphine; Randomised clinical trial
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Morphine (Experimental): 2.5 mg dose of epidural morphine given within one hour following vaginal delivery
  Interventions: Drug: Preservative-free epidural morphine
- Placebo (Placebo Comparator): 5 ml of epidural preservative-free saline given within one hour following vaginal delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Preservative-free epidural morphine — One time dose of preservative-free epidural morphine 2.5 mg given within one hour following vaginal delivery
  Other Names: Morphine; Epidural Narcotics
  Arms: Epidural Morphine
Drug: Placebo — 5 ml of epidural preservative-free saline given within one hour following vaginal delivery
  Arms: Placebo

SUMMARY:
The investigators believe that pain management following a vaginal delivery can be improved. Many women receive epidural medication during labor and delivery, and the investigators felt that using the epidural following delivery might improve the first day pain. This study is to determine whether a single dose of epidural morphine given to mothers after a vaginal delivery will reduce the perineal pain in the postpartum period.

DETAILED DESCRIPTION:
Vaginal deliveries comprise 80-85% of all deliveries. Although this is felt to be natural and safe, this route can be associated with significant perineal trauma and subsequent postpartum perineal pain. The degree of perineal trauma varies from the minimum of vaginal stretching and distension associated with labor, to episiotomy and significant perineal tears. In spite of the differences in the degree of injury following vaginal delivery, postpartum pain therapy is poorly organized and at best consists of simple analgesics and anti-inflammatory drugs. The purpose of this study is to determine if a single dose of epidural-administered morphine offers additional advantage to an organized program for the management of immediate postpartum perineal pain following vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients (ASA 1 or 2) of > 34 weeks gestational age who chose epidural analgesia for labor, and deliver vaginally.

Exclusion Criteria:

* Women whose labor is terminated by cesarean delivery
* Parturients with known morphine allergy
* Parturients with narcotic addiction past / present

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 228 (Actual)
Dates: Start 2002-03; Primary Completion 2004-11 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Macarthur, MD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Goodman SR, Drachenberg AM, Johnson SA, Negron MA, Kim-Lo SH, Smiley RM. Decreased postpartum use of oral pain medication after a single dose of epidural morphine. Reg Anesth Pain Med. 2005 Mar-Apr;30(2):134-9. doi: 10.1016/j.rapm.2004.11.010. PMID 15765455
- [Background] Macdonald R, Smith PJ. Extradural morphine and pain relief following episiotomy. Br J Anaesth. 1984 Nov;56(11):1201-5. doi: 10.1093/bja/56.11.1201. PMID 6386019
- [Background] Niv D, Wolman I, Yashar T, Varrassi G, Rudick V, Geller E. Epidural morphine pretreatment for postepisiotomy pain. Clin J Pain. 1994 Dec;10(4):319-23. doi: 10.1097/00002508-199412000-00013. PMID 7858363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parturients were recruited at Mount Sinai Hospital labor and delivery unit. Recruitment took place between March 2002 and November 2004.
Pre-assignment Details: Parturients were approached prior to delivery if they had received epidural analgesia for labor. Following a vaginal delivery, the subject was randomized to one of the two arms.
Period: Overall Study
Arm/Group | Epidural Morphine | Placebo
Started | 113 | 115
Completed | 113 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Morphine | Placebo | Total
Number analyzed (Participants) | 113 | 115 | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (4.9) | 31.8 (4.9) | 32.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 115 | 228
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Number of caucasian, non-caucasian study subjects
  Participants
    Caucasian | 87 | 99 | 186
    Non-caucasian | 17 | 11 | 28
    Missing information | 9 | 5 | 14
Operative vaginal delivery [Number; unit: participants] — Number of study subjects with spontaneous, operative vaginal delivery
  participants
    Operative vaginal delivery | 38 | 34 | 72
    Spontaneous vaginal delivery | 75 | 81 | 156
Parity [Number; unit: participants] — Number of primiparous, multiparous study subjects
  participants
    Primiparous | 76 | 79 | 155
    Multiparous | 37 | 36 | 73
Perineal Trauma [Number; unit: Participants] — Number of subjects with minimal, major perineal tears
  Participants
    Second degree tear or greater | 82 | 87 | 169
    First degree tear or less | 31 | 28 | 59
Maternal Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.0 (5.9) | 29.0 (6.6) | 29.0 (6.2)
Neonatal Birth Weight [Mean (Standard Deviation); unit: kilograms] | 3.4 (0.51) | 3.4 (0.46) | 3.4 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Women Who Received Systemic Narcotic Analgesics in the First 24 Hours Postpartum
Time Frame: 24 hours postpartum
Population: Analysis by intention to treat.
Measure: Number; unit: participants
Arm/Group | Epidural Morphine | Placebo
Number analyzed (Participants) | 113 | 115
participants | 8 | 37
Statistical Analysis 1: Comparison: Epidural Morphine vs Placebo; Relative risk ratio estimation with 95% CI using exact methods; Test type: Superiority or Other; p = 0.05, Fisher Exact; Risk Ratio (RR) = 0.22, 95% CI [0.12 to 0.41] — Relative risk describes the risk of requiring additional analgesics in the first 24 hours postpartum with the denominator being the arm which received placebo

2. Secondary Outcome: Time to First Request for Analgesia
Description: All participants requested analgesia at least once during their hospitalization
Time Frame: Hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Epidural Morphine | Placebo
Number analyzed (Participants) | 113 | 115
hours | 22.9 (4.0) | 18.9 (8.0)
Statistical Analysis 1: Comparison: Epidural Morphine vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; degrees of freedom 226; Mean Difference (Final Values) = -4.0, 95% CI [-5.7 to -2.3], Standard Error of Mean 0.8 — The epidural morphine group represents the baseline of comparison for difference in means, with the placebo group requiring additional analgesics earlier

3. Secondary Outcome: Maternal Visual Analogue Scale (VAS) Score at Time of Request for First Additional Analgesic
Description: Participants were asked to indicate on a 10 cm line the point at which their perineal pain scored between one end anchored with "no pain in my bottom" to the other end anchored with "the worst pain in my bottom that I can imagine"
Time Frame: by 24 hours postpartum
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Epidural Morphine | Placebo
Number analyzed (Participants) | 113 | 115
scores on a scale | 0.3 (1.4) | 1.6 (2.7)
Statistical Analysis 1: Comparison: Epidural Morphine vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; degrees of freedom 212; Mean Difference (Final Values) = 1.3, 95% CI [0.7 to 1.8], Standard Error of Mean 0.3 — Difference in VAS score when compared to the baseline group, subjects receiving epidural morphine

4. Secondary Outcome: Maternal Satisfaction With Perineal Pain Management
Description: 5 point Likert scale asking for agreement with the statement "I was satisfied with my pain relief for the pain in my bottom during the first day after delivery". Scale ranged from strongly disagree to strongly agree.
Time Frame: at 24 hours postpartum
Measure: Number; unit: participants
Arm/Group | Epidural Morphine | Placebo
Number analyzed (Participants) | 113 | 115
participants
  Strongly Disagree | 1 | 3
  Disagree | 9 | 11
  Not sure | 6 | 8
  Agree | 43 | 38
  Strongly Agree | 45 | 45
  Missing information | 9 | 10
Statistical Analysis 1: Comparison: Epidural Morphine vs Placebo; Test type: Superiority or Other; p = 0.80, Fisher Exact — Fisher's exact test result did not reveal statistically significant differences between expected and real frequencies in any of the categories

5. Secondary Outcome: Side Effects
Description: Number of participants with pruritus, nausea and vomiting, urinary retention, drowsiness in the first 24 hours postpartum
Time Frame: at 24 hours postpartum
Reporting Status: Not Posted
Measure: Number; unit: Number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No